CLINICAL TRIAL: NCT02349048
Title: A Phase 2, Randomized, Open-label Study to Investigate the Efficacy, Safety, Tolerability and Pharmacokinetics of 6 or 8 Weeks of Treatment With Simeprevir, Daclatasvir and Sofosbuvir in Treatment-naive Subjects With Chronic Hepatitis C Virus Genotype 1 Infection
Brief Title: Study to Assess Efficacy, Safety, Tolerability and Pharmacokinetics of Simeprevir, Daclatasvir and Sofosbuvir in Treatment-naive Participants With Chronic Hepatitis C Virus Genotype 1 Infection
Acronym: ACCORDION-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR105963; TMC435HPC2013 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C virus; Hepatitis C virus genotype 1; Chronic Hepatitis C Virus Genotype 1 Infection; Liver fibrosis; Cirrhosis; Simeprevir; Daclatasvir; Sofosbuvir
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis; Fibrosis | interventions — Simeprevir; daclatasvir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Chronic hepatitis C virus (HCV) genotype 1 infected participants with early stages of liver fibrosis, will receive Simeprevir (SMV) 150 milligram (mg), Daclatasvir (DCV) 60 mg and Sofosbuvir (SOF) 400 mg once daily for 6 weeks.
  Interventions: Drug: Simeprevir 150 mg; Drug: Daclatasvir 60 mg; Drug: Sofosbuvir 400 mg
- Arm B (Experimental): Chronic HCV genotype 1 infected participants with cirrhosis, will receive SMV 150 mg, DCV 60 mg and SOF 400 mg once daily for 8 weeks.
  Interventions: Drug: Simeprevir 150 mg; Drug: Daclatasvir 60 mg; Drug: Sofosbuvir 400 mg

INTERVENTIONS:
Drug: Simeprevir 150 mg — Simeprevir 150 mg capsule orally once daily.
Drug: Daclatasvir 60 mg — Daclatasvir 60 mg tablet orally once daily.
Drug: Sofosbuvir 400 mg — Sofosbuvir 400 mg tablet orally once daily.

SUMMARY:
The purpose of this study is to evaluate the efficacy of 6 or 8 weeks of treatment regimen containing simeprevir (SMV), daclatasvir (DCV) and sofosbuvir (SOF) in treatment-naive (not having received treatment with any approved or investigational drug) participants with chronic hepatitis (inflammation of the liver) C virus (HCV) genotype 1 infection with early stages of liver fibrosis or with cirrhosis.

DETAILED DESCRIPTION:
This is an open-label (participants and researchers are aware about the treatment participants are receiving), and multicenter (when more than 1 hospital or medical school team work on a medical research) study. The study will consist of a Screening Phase (6 weeks); an Open-label Treatment Phase (6 weeks for Arm A and 8 weeks for Arm B); and a Post-treatment Follow-up Phase (until 24 weeks after end of study treatment). Using a staggered approach, all eligible participants will be assigned to 1 of the 2 arms, according to their level of fibrosis. Arm A (consists of chronic HCV genotype 1 infected participants with early stages of liver fibrosis): participants will receive a combination therapy of SMV 150 milligram (mg), DCV 60 mg and SOF 400 mg once daily for 6 weeks. Arm B (consists of chronic HCV genotype 1 infected participants with cirrhosis): participants will receive a combination therapy of SMV 150 mg, DCV 60 mg and SOF 400 mg once daily for 8 weeks. A sub-study will be performed at a selected study site, where only participants who will be eligible to participate in both the main study and the sub-study will be enrolled. Intra-hepatic and plasma HCV ribonucleic acid (RNA) levels; intra-hepatic, peripheral innate and adaptive immune responses during the treatment, will be assessed in the sub-study. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* HCV genotype 1 infection and HCV RNA plasma level greater than (>) 10,000 international units per milliliter (IU/mL), both determined at Screening
* Participants of Arm A should have evidence of early stages of liver fibrosis, defined by a FibroSURE score less than or equal to (<=) 0.48 and aspartate aminotransferase to platelet ratio index (APRI) score <=1
* Participants of Arm B should have evidence of cirrhosis, defined by a FibroSURE score >0.75 and APRI score >2, OR a previous (historical) biopsy documenting a METAVIR score F4. In addition, participants should have absence of esophageal varices or presence of small (grade 1) esophageal varices determined by upper gastrointestinal endoscopy, and absence of findings indicative of hepatocellular carcinoma in an ultrasonography
* HCV treatment-naive, defined as not having received treatment with any approved or investigational drug for chronic HCV infection
* Pegylated interferon (PegIFN) and ribavirin (RBV) eligible, defined as not having any contraindication to the use of PegIFN and RBV, in line with the prescribing information for each compound

Exclusion Criteria:

A. Main Study:

* Co-infection with HCV of another genotype than genotype 1 and/or human immunodeficiency virus (HIV) type 1 or 2 (positive HIV-1 or HIV 2 antibody test at Screening)
* Any evidence of liver disease of non-HCV etiology. This includes, but is not limited to, acute hepatitis A infection, hepatitis B infection (hepatitis B surface antigen positive), drug- or alcohol-related liver disease, autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, non-alcoholic steatohepatitis, primary biliary cirrhosis, or any other non-HCV liver disease considered clinically significant by the Investigator
* Evidence of clinical hepatic decompensation or presence of grade 2/3 esophageal varices
* Any of the protocol defined laboratory abnormalities

B. Sub-study:

* Presence of coagulopathy (hemophilia) or hemoglobinopathy (including sickle cell disease, thalassemia)
* Use of any anti-coagulant (for example, warfarin, heparin) or anti-platelet medications within 1 week of the Screening visit
* Any of the protocol defined laboratory abnormalities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- United States (7):
  - Bakersfield, California
  - Jacksonville, Florida
  - Lutherville, Maryland
  - Winston-Salem, North Carolina
  - Knoxville, Tennessee
  - Arlington, Texas
  - San Antonio, Texas
- Toronto, Ontario, Canada

REFERENCES:
- [Derived] Sulkowski MS, Feld JJ, Lawitz E, Felizarta F, Corregidor AM, Khalid O, Ghalib R, Smith WB, Van Eygen V, Luo D, Vijgen L, Gamil M, Kakuda TN, Ouwerkerk-Mahadevan S, Van Remoortere P, Beumont M. Efficacy and safety of 6 or 8 weeks of simeprevir, daclatasvir, sofosbuvir for HCV genotype 1 infection. J Viral Hepat. 2018 Jun;25(6):631-639. doi: 10.1111/jvh.12853. Epub 2018 Feb 6. PMID 29274193

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks: Chronic hepatitis C virus (HCV) genotype 1 infected participants with early stages of liver fibrosis received therapy (Simeprevir [SMV] 150 milligram (mg)/Daclatasvir [DCV] 60mg/Sofosbuvir [SOF] 400mg) once daily for 6 weeks.
- Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks: Chronic hepatitis C virus (HCV) genotype 1 infected participants with compensated cirrhosis received therapy (Simeprevir [SMV] 150 milligram (mg)/Daclatasvir [DCV] 60mg/Sofosbuvir [SOF] 400mg) once daily for 8 weeks.
Period: Overall Study
Arm/Group | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks
Started | 59 | 9
Completed | 54 | 9
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks | Total
Number analyzed (Participants) | 59 | 9 | 68
Age, Continuous [Median (Full Range); unit: years] | 47 [18 to 63] | 56 [52 to 64] | 50.5 [18 to 64]
Gender [Count of Participants; unit: Participants]
  Female | 32 | 5 | 37
  Male | 27 | 4 | 31
Region of Enrollment [Number; unit: participants]
  CAN | 9 | 0 | 9
  USA | 50 | 9 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After End of Study Drug Treatment (SVR12)
Description: Participants were considered to have achieved SVR12 if the hepatitis C virus ribonucleic acid (HCV RNA) was less than (<) lower limit of quantification (LLOQ; 15 international unit per milliliter [IU/mL]) detectable or undetectable at 12 weeks after the end of study drug treatment.
Time Frame: 12 weeks after end of study drug treatment (week 18 for Arm A and week 20 for Arm B)
Population: The Intent-to-treat (ITT) analysis set is defined as all enrolled participants who took at least 1 dose of Simeprevir (SMV), Sofosbuvir (SOF) or Daclatasvir (DCV).
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks
Number analyzed (Participants) | 59 | 9
Percentage of Participants | 86.4 | 100

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Response
Description: On-treatment virologic response was determined by hepatitis C virus (HCV) ribonucleic acid (RNA) results satisfying a specified threshold.
  The following thresholds were considered at any time point: <LLOQ undetectable, <LLOQ detectable, and <LLOQ undetectable or detectable. The LLOQ value was 15 IU/mL. Very rapid virologic response (vRVR) is undetectable HCV RNA at Week 2 while on treatment and Rapid virologic response (RVR) is undetectable HCV RNA at Week 4 while on treatment.
Time Frame: Day 2, Day 3, Week 1, 2, 3, 4, 6 (for Arm A) and 8 (for Arm B only)
Population: The Intent-to-treat (ITT) analysis set is defined as all enrolled participants who took at least 1 dose of Simeprevir (SMV), Sofosbuvir (SOF) or Daclatasvir (DCV). Here 'n' signifies number of participants who were evaluable at each specified time point, for each arm, respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks
Number analyzed (Participants) | 59 | 9
Percentage of Participants
  Day 2 : >= 15 IU/mL (n = 56, 9) | 96.4 | 100
  Day 2 : < 100 IU/mL (n = 56, 9) | 7.1 | 0
  Day 2 : < 15 IU/mL undetect/detectable (n = 56, 9) | 3.6 | 0
  Day 2 : < 15 IU/mL detectable (n = 56, 9) | 3.6 | 0
  Day 2: < 15 IU/mL undetectable (n = 56, 9) | 0 | 0
  Day 3 : >= 15 IU/mL (n = 58, 9) | 94.8 | 100
  Day 3 : < 100 IU/mL (n = 58, 9) | 19.0 | 11.1
  Day 3 : < 15 IU/mL undetect/detectable (n = 58, 9) | 5.2 | 0
  Day 3 : < 15 IU/mL detectable (n = 58, 9) | 5.2 | 0
  Day 3 : < 15 IU/mL undetectable (n = 58, 9) | 0 | 0
  Week 1: >= 15 IU/mL (n = 58, 9) | 58.6 | 66.7
  Week 1: < 100 IU/mL (n = 58, 9) | 75.9 | 33.3
  Week 1: < 15 IU/mL undetect/detectable (n = 58, 9) | 41.4 | 33.3
  Week 1 : < 15 IU/mL detectable (n = 58, 9) | 36.2 | 33.3
  Week 1 : < 15 IU/mL undetectable (n = 58, 9) | 5.2 | 0
  Week 2 : >= 15 IU/mL (n = 56, 9) | 19.6 | 66.7
  Week 2: < 100 IU/mL (n = 56, 9) | 94.6 | 77.8
  Week 2: < 15 IU/mL undetect/detectable (n = 56, 9) | 80.4 | 33.3
  Week 2 : < 15 IU/mL detectable (n = 56, 9) | 41.1 | 0
  Week 2: < 15 IU/mL undetectable (vRVR) (n = 56, 9) | 39.3 | 33.3
  Week 3: >= 15 IU/mL (n = 56, 9) | 7.1 | 33.3
  Week 3: < 100 IU/mL (n = 56, 9) | 100 | 100
  Week 3: < 15 IU/mL undetect/detectable (n = 56, 9) | 92.9 | 66.7
  Week 3 : < 15 IU/mL detectable (n = 56, 9) | 21.4 | 22.2
  Week 3 : < 15 IU/mL undetectable (n = 56, 9) | 71.4 | 44.4
  Week 4 : >= 15 IU/mL (n = 58, 9) | 3.4 | 11.1
  Week 4: < 100 IU/mL (n = 58, 9) | 98.3 | 100
  Week 4: < 15 IU/mL undetect/detectable (n = 58, 9) | 96.6 | 88.9
  Week 4 : < 15 IU/mL detectable ( n = 58, 9) | 8.6 | 33.3
  Week 4 : < 15 IU/mL undetectable (RVR) (n = 58, 9) | 87.9 | 55.6
  Week 6 : >= 15 IU/mL (n = 58, 9) | 0 | 0
  Week 6: < 100 IU/mL ( n = 58, 9) | 100 | 100
  Week 6: < 15 IU/mL undetect/detectable (n = 58, 9) | 100 | 100
  Week 6 : < 15 IU/mL detectable (n = 58, 9) | 6.9 | 0
  Week 6 : < 15 IU/mL undetectable (n= 58, 9) | 93.1 | 100
  Week 8 : >= 15 IU/ml (n = 0, 9) | NA — HCV RNA values were not collected at week 8 since participants in Arm A ended treatment at week 6. | 0
  Week 8: < 100 IU/mL (n = 0, 9) | NA — HCV RNA values were not collected at week 8 since participants in Arm A ended treatment at week 6. | 100
  Week 8: < 15 IU/mL undetect/detectable (n = 0, 9) | NA — HCV RNA values were not collected at week 8 since participants in Arm A ended treatment at week 6. | 100
  Week 8: < 15 IU/mL detectable (n = 0, 9) | NA — HCV RNA values were not collected at week 8 since participants in Arm A ended treatment at week 6. | 0
  Week 8: < 15 IU/mL undetectable (n = 0, 9) | NA — HCV RNA values were not collected at week 8 since participants in Arm A ended treatment at week 6. | 100

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 Weeks (SVR4) and 24 Weeks (SVR24) After End of Study Drug Treatment
Description: Participants were considered to have achieved SVR4 and SVR24 if the HCV RNA was <LLOQ detectable or undetectable at 4 weeks and 24 weeks respectively after the end of study drug treatment. The LLOQ value was 15 IU/mL.
Time Frame: 4 weeks after end of study drug treatment (week 10 for Arm A and 12 for Arm B); 24 weeks after end of study drug treatment (week 30 for Arm A and 32 for Arm B)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks
Number analyzed (Participants) | 59 | 9
Percentage of Participants
  SVR4 | 93.2 | 100
  SVR24 | 84.7 | 100

4. Secondary Outcome: Percentage of Participants With On-Treatment Failure
Description: Participants who did not achieve SVR12 and with confirmed detectable HCV RNA at the actual end of treatment. Includes participants with: 1) viral breakthrough, defined as a confirmed increase of greater than (>)1 log10 in HCV RNA from nadir, or confirmed HCV RNA 2) confirmed detectable HCV RNA at the actual end of treatment (example, completed treatment, discontinued due to adverse events, withdrawal of consent) of >100 IU/mL in participants whose HCV RNA had previously been <LLOQ while on treatment.
Time Frame: Baseline up to End of Treatment (Week 6 for Arm A and Week 8 for Arm B)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks
Number analyzed (Participants) | 59 | 9
Percentage of Participants | 1.7 | 0

5. Secondary Outcome: Number of Participants With Viral Relapse
Description: Viral Relapse: Participants who did not achieve SVR12, with undetectable HCV RNA at the actual end of study drug treatment and confirmed HCV RNA greater than or equal to (>=) LLOQ during followup.
Time Frame: From Week 6 to Week 18 (for Arm A) and From Week 8 to Week 20 (for Arm B)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks
Number analyzed (Participants) | 59 | 9
Participants | 7 | 0

6. Secondary Outcome: Number of Participants With Late Viral Relapse
Description: Late Viral Relapse: Participant who achieved SVR12 and the post treatment HCV RNA measurement fulfilled 1 the following conditions: a) at least 2 consecutive measurements not lesser than (<)15 IU/mL undetectable, of which at least the second measurement was >=15 IU/mL quantifiable or b) the last available measurement was >=15 IU/mL quantifiable.
Time Frame: From Week 18 to Week 30 (for Arm A), From Week 20 to Week 32 (for Arm B)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks
Number analyzed (Participants) | 59 | 9
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With HCV Nonstructural Protein 3/4A (NS3/4A), NS5A and NS5B Sequence in Participants Not Achieving SVR
Description: Sequencing of the HCV nonstructural protein 3/4A (NS3/4A), nonstructural protein 5A (NS5A) and nonstructural protein 5B (NS5B) genes was done to identify preexisting sequence polymorphisms and characterize emerging HCV viral variants in participants not achieving SVR.
Time Frame: Up to Week 30 for Arm A and up to Week 32 for Arm B
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks
Number analyzed (Participants) | 59 | 9
Participants | 8 | 0

8. Secondary Outcome: Percentage of Participants With or Without an NS3 Q80K Polymorphism at Baseline Achieving SVR
Description: The Q80K polymorphism, associated with low level SMV in vitro resistance. Percentage of participants who achieved SVR with or without an NS3 Q80K polymorphism at baseline were reported.
Time Frame: up to Week 30 for Arm A and Week 32 for Arm B
Population: The ITT analysis set is defined as all enrolled participants who took at least 1 dose of SMV, SOF or DCV. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' signifies number of participants evaluable for this outcome measure at specific time point.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks
Number analyzed (Participants) | 25 | 9
Percentage of Participants
  With NS3 Q80K polymorphism at baseline (n=25,9) | 88.0 | 100
  Without NS3 Q80K polymorphism at baseline (n=23,9) | 78.3 | 100

ADVERSE EVENTS:
Time Frame: Only adverse events from the Treatment Period (6 weeks in Arm A and 8 weeks in Arm B) are reported.
Arm/Group | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks
Serious Adverse Events (participants affected / at risk) | 1/59 | 0/9
Other Adverse Events (participants affected / at risk) | 39/59 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks (N=59) | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks (N=9)
Chest Pain (General disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Simeprevir/Daclatasvir/Sofosbuvir - 6 Weeks (N=59) | Arm B: Simeprevir/Daclatasvir/Sofosbuvir - 8 Weeks (N=9)
Cataract (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 1
Fatigue (General disorders) | 14 | 1
Nasopharyngitis (Infections and infestations) | 4 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 6 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 15 | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The sample size in Arm B (participants with cirrhosis) was small (n=9).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.